CLINICAL TRIAL: NCT05427734
Title: Drivers of Suicide Mobile App Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Evidence-Based Practice Institute, Seattle, WA (Industry)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R44AA029868 (NIH); R44AA029868 (NIH)
Record Dates: First submitted 2022-06-15; First posted 2022-06-22 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Suicide; Suicide, Attempted; Suicidal Ideation; Alcohol Use Disorder; Alcoholism; Alcohol Abuse; Screening and Brief Interventions
MeSH Terms: conditions — Suicide; Suicide, Attempted; Suicidal Ideation; Alcoholism

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (2):
- WisePath for Adults (Experimental): WisePath is designed to help support individuals during challenging moments and while experiencing behavioral concerns. The app is designed for people who struggle with depression, sleep problems, have feelings of wanting to die, or want to harm themselves, and/or misuse alcohol. WisePath includes specific tools for those who are experiencing suicidality, including creating a safety plan and teaching skills and strategies to get through distressing moments. You have been assigned to use the WisePath app while you are in this study.
  Interventions: Device: WisePath for Adults
- Active-Control app + electronic wellness resources brochure (Active Comparator): Well-regarded suicide prevention self-help app, plus an electronic wellness resources brochure containing links to health and wellness materials, psychoeducation about suicide, depression, self-help recovery-focused resources (e.g., Alcoholics Anonymous, other 12-Step programs, Moderation Management, etc.), and phone/text information for the National Suicide Prevention Lifeline.
  Interventions: Device: Active-Control app + electronic wellness resources brochure

INTERVENTIONS:
Device: WisePath for Adults — Participants assigned to this condition will receive access to the WisePath app for 12 weeks.
  Arms: WisePath for Adults
Device: Active-Control app + electronic wellness resources brochure — Participants assigned to this condition will receive access to Virtual Hope Box, a well-regarded suicide prevention self-help app, for 12 weeks plus an electronic wellness resources brochure.
  Arms: Active-Control app + electronic wellness resources brochure

SUMMARY:
The central purpose of this project is to evaluate and facilitate access to evidence-based best practices for individuals struggling with suicidal ideation and co-occurring behavioral problems, including alcohol misuse, and provide assistance to the patients while they are waiting to receive care, as they are receiving care, and after they return home. While WisePath is highly innovative in how it delivers these best practices, the content is well-established and known to reduce suicidality and alcohol misuse.

We will conduct a 12-week intent-to-treat RCT with 120 suicidal adults 22 years and older who may also be experiencing alcohol misuse. Participants will be randomly assigned to WisePath (n=60) or an active control condition (n=60) including a control suicide prevention self-help app plus an electronic wellness resources brochure containing links to health and wellness materials, psychoeducation about suicide, depression, self-help recovery-focused resources (e.g., Alcoholics Anonymous and other 12-Step programs, Moderation Management, etc.), and phone/text information for the 988 Suicide & Crisis Lifeline. Participants will be assessed at baseline, 4, 8 and 12 weeks.

DETAILED DESCRIPTION:
This study will test the newly developed WisePath for Adults ("WisePath"), a robust digital technology developed under NIAAA SBIR Fast-Track award (R44AA029868; Drs. Dimeff & Jobes, Co-PIs) that is developed to efficiently and reliably aid delivery of recommended best-practices for the treatment of suicidal ideation in adults, including suicidal individuals who also misuse alcohol. WisePath includes techniques for prevention of suicidal behaviors (ideation, planning, attempts) while providing access to support resources in the moment via a mobile app. WisePath will include evidence-based practices for suicide prevention, including for those who are suicidal and also experience other behavioral health concerns such as depressed mood, sleep problems, and misuse of alcohol. This study will test WisePath with individuals who are experiencing these problems and recently sought treatment from a primary care provider. WisePath includes: psychoeducation, behavioral skills training, crisis stabilization planning, lethal means management, brief interventions for the treatment of suicidal ideation, depressed mood, sleep problems, alcohol misuse, and messages of hope, wisdom, and insights from people with lived experience (PLE).

We will conduct a randomized controlled trial (RCT; N=120) comparing WisePath (n=60) to an active control condition (a well-regarded suicide prevention self-help app + electronic wellness resources brochure; n=60) in adults experiencing suicidal ideation. To ensure a sufficient sample of individuals who misuse alcohol, no fewer than 35% (n=42) of the sample will be comprised of individuals who experience a harmful or hazardous level of alcohol use. Participants will be randomly assigned to a condition utilizing a minimization randomization procedure to match participants across condition on suicide severity, depression severity, and alcohol misuse. Participants will be assessed at baseline, 4, 8, and 12 weeks.

We hypothesize that in comparison to the active control condition, WisePath participants will show significantly better outcomes from baseline to the 4-, 8-, and 12-week assessment points such that:

1. WisePath participants will report significantly greater decreases in suicidal and alcohol misuse behaviors compared to controls
2. WisePath participants will report greater increases in self-efficacy and coping with suicidal thoughts and distress, as well as use of suicide prevention strategies compared to study controls
3. WisePath participants will report a higher degree of satisfaction with their respective app compared to controls

ELIGIBILITY:
Inclusion Criteria:

* Resides in the United States
* 22+ years of age
* English speaking
* At risk for suicide, as evidenced by at least one of the following:
* One or more lifetime suicide attempts (ASQ item 4)
* Endorsement of any ASQ items 1 -3 (expanded from "past few weeks" in ASQ to "past 30 days" in our measures)

  * Item 1: In the past 30 days, have you wished you were dead?
  * Item 2: In the past 30 days, have you felt that you or your family would be better off if you were dead?
  * Item 3: In the 30 days, have you been having thoughts about killing yourself?
* Currently has a primary care provider and sought care from them in the past year
* Possesses and is the primary user of an Android- or iPhone-based smartphone with a data plan

Given that alcohol misuse exponentially increases the risk of death by suicide, can exacerbate other problems, and interfere with effective treatment, we will over-recruit individuals who misuse alcohol to ensure relevance of the tool for them. No fewer than 35% of the sample will be comprised of individuals who score 8 or more on the Alcohol Use Disorders Identification Test (AUDIT), indicating a harmful or hazardous level of drinking.

To ensure a sufficient sample of individuals who misuse alcohol, no fewer than 35% of the sample will be comprised of individuals who score 8 or more on the Alcohol Use Disorders Identification Test (AUDIT), indicating a harmful or hazardous level of drinking.

Exclusion Criteria:

* Severe depression (PHQ-9 score of 20 or greater)
* Alcohol dependence (AUDIT score of 32 or greater)
* Acutely suicidal (affirms item 5 of the Ask Suicide Screening Questions; Are you having thoughts of killing yourself right now? Followed by endorsing intent; Have you intended to act on urges to kill yourself in the past 30 days? or planning within the past 30 days; Have you made a plan to kill yourself in the past 30 days?)
* Significant drug abuse problems (scores 6 or greater on the DAST-10)

Individuals who are excluded because of the severity of their depression, suicide acuity, and/or degree of substance use disorder will be provided with resources (i.e., the Suicide and Crisis Lifeline (988), SAMHSA's National Helpline) and encouraged to reach out to their primary care or mental/behavioral health provider.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2025-03-05 (Actual); Primary Completion 2025-11-10 (Actual); Study Completion 2025-11-10 (Actual)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire-9 | Eligibility Screening (time 0), 4 weeks (time 2), 8 weeks (time 3), 12 weeks (time 4)
  9-item self-report measure (minimum of 0 and maximum of 27) that assesses recent depressive symptoms, and has excellent sensitivity (.77 to .86) and specificity (.78 to .95) in detecting major depression. Scores of 1-9 indicate minimal to mild depression; 10-14, moderate depression; 15-19, moderately severe depression; and 20-27, severe depression.
Change in Self-Injurious Thoughts and Behaviors Interview-Revised | Baseline (time 1), 4 weeks (time 2), 8 weeks (time 3), 12 weeks (time 4)
  A structured interview, which can also be delivered as a self-report measure, containing modules that assess suicidal ideation, suicide plans, suicide gestures, suicide attempts, and non-suicidal self injury. The SITBI has excellent psychometric properties, with inter-rater reliability coefficients in the range of 1.0 and strong test-retest reliability over six months. The SITBI correlates highly and in expected directions with other suicidal ideation measures and is behaviorally specific.
Change in Suicide-Related Coping Scale | Baseline (time 1), 4 weeks (time 2), 8 weeks (time 3), 12 weeks (time 4)
  17-item psychometrically-sound self-report measure (minimum of 0 and maximum of 68) of coping with suicidal thoughts, urges, and crises that uses a 5-point rating scale (0=strongly disagree; 4=strongly agree). Higher scores indicate higher ability to cope with suicidality.
Change in the Patient-Reported Outcome Measurement Information System (PROMIS) | Baseline (time 1), 4 weeks (time 2), 8 weeks (time 3), 12 weeks (time 4)
  A well-validated, normed set of measures with standardized scoring. All measures are scored on a 5-point scale and responses are summed to create a raw total score for each measure. The raw scores are then rescaled to T-scores with a mean of 50 and standard deviation of 10.

SECONDARY OUTCOMES:
Change in Suicide Attempt Self-Injury Interview | Baseline (time 1), 4 weeks (time 2), 8 weeks (time 3), 12 weeks (time 4)
  A gold-standard interviewer-administered instrument used to gather information about the occurrence of suicidal and NSSI, including the frequency, intent, medical severity, outcomes for each event during the assessment window, as well as healthcare utilization associated with suicidal behavior. Includes a six-item self-report measure assessing frequency of engagement in suicidal or self-injurious behaviors as well as the frequency of seeking assistance from emergency room, professional, or crisis line for suicidal or self-injurious behaviors in the past three months.
App Satisfaction Survey | 12 weeks (time 4)
  An eight-item survey used in EBPI's earlier research, which focuses on an app's ease of use and helpfulness. The initial six items use a five-point rating scale (1=poor; 5=excellent). Users also provide an overall satisfaction rating for their condition app using a 100-point scale and indicate whether they would recommend using the app to others in their situation.

OTHER OUTCOMES:
Demographics Questionnaire | Eligibility Screening (time 0)
  Self-report measure to collect demographics from participants in this study. Questions include items about gender, race, and ethnicity.
Ask Suicide Screening Questions | Eligibility Screening (time 0)
  A five-item brief validated screening tool for youth and adults and developed by NIMH researchers to help healthcare providers identify individuals at risk for suicide. ASQ Item 5 assesses immediate acuity of suicidality. All items are yes or no questions.
Alcohol Use Disorders Identification Test | Eligibility Screening (time 0)
  10-item psychometrically sound self-report measure (minimum of 0 and maximum of 40) used in a variety of healthcare settings worldwide to assess alcohol intake, potential dependence on alcohol, and experience of alcohol-related harm. Scores from 8 to 15 suggest hazardous or harmful alcohol consumption and a score of 16 or more indicates the likelihood of alcohol dependence (moderate-severe alcohol use disorder).
Drug Abuse Screening Test | Eligibility Screening (time 0)
  10-item psychometrically validated self-administered screening tool for drug-related problems. Each question answered "yes" is scored as 1 point (question 3 is reverse-scored) and total is summed where 0 is no problems reported through 10, severe level of problems related to drug abuse.
Columbia-Suicide Severity Rating Scale | Eligibility Screening (time 0)
  A FDA-recommended tool to assess suicidal behaviors in healthcare systems. Investigators will use the C-SSRS items to assess suicide attempts for purposes of the eligibility screening. It contains 6 yes or no questions.
Eligibility Screen | Eligibility Screening (Time 0)
  Brief survey conducted prior to consent to help determine if individual is eligible for the study.

CONTACTS AND LOCATIONS:
Overall Officials: Linda A. Dimeff, PhD, Principal Investigator — Chief Executive Officer
Locations (1):
- Evidence-Based Practice Institute, Inc., Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Requests for use of data will be considered on a case-by-case basis. Interested researchers may send data requests to research@jasprhealth.com.
  The final dataset will include self-reported demographic and behavioral data from participants in the randomized controlled trial. The dataset will include sensitive data from participants regarding suicidal behavior and substance use. Even though the final dataset will be stripped of identifiers prior to release for sharing, investigators believe that there remains the possibility of deductive disclosure of participants. Thus, the de-identified dataset will be distributed by Drs. Dimeff and Jobes to those that request it and only under a data-sharing agreement that includes: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate security protections; and (3) a commitment to destroying the data after analyses are completed.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Study data will become available after grant closeout, in perpetuity.
Access Criteria: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate security protections; and (3) a commitment to destroying the data after analyses are completed.